CLINICAL TRIAL: NCT04258553
Title: Evaluation of Thiol Disulfide Balance in Cervix Cancer
Brief Title: Thiol Disulfide Balance in Cervix Cancer
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Burak Sezgin, Principal Investigator, Muğla Sıtkı Koçman University
Other Study IDs: 19/09/2018-15-4
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Cervix Cancer; Oxidative Stress
Keywords: thiol disulfide hemostasis; screening; early diagnosis
MeSH Terms: conditions — Uterine Cervical Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum blood samples for each participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cervix cancer: Cervix cancer n=62
  Interventions: Diagnostic Test: Disulphide(μmol/L); Diagnostic Test: Total Oxidant Capacity(μmolH2O2Equiv/L); Diagnostic Test: Ischemia Modified Albumin(IU/mL)
- Healthy controls: Healthy volunteers n=61
  Interventions: Diagnostic Test: Disulphide(μmol/L); Diagnostic Test: Total Oxidant Capacity(μmolH2O2Equiv/L); Diagnostic Test: Ischemia Modified Albumin(IU/mL)

INTERVENTIONS:
Diagnostic Test: Disulphide(μmol/L) — Aforementioned oxidative stress markers will be measured via Cobas c501(Roche Diagnostics, Indianapolis, IN, USA) used with spectrophotometry
  Other Names: Native thiol (μmol/L); Total thiol (μmol/L); Native thiol/totalthiol(%); Disulfide/native thiol(%); Disulfide/total thiol(%)
Diagnostic Test: Total Oxidant Capacity(μmolH2O2Equiv/L) — Aforementioned oxidative stress markers will be measured via Cobas c501(Roche Diagnostics, Indianapolis, IN, USA) used with spectrophotometry
  Other Names: Total Antioxidant Capacity(mmolTroloxEquiv/L); Oxidative stress Index (Arbitrary Unite)
Diagnostic Test: Ischemia Modified Albumin(IU/mL) — The serum Ischemia Modified Albumin concentrations were measured as described by Bar-Or et al. (Bar-Or et al. 2000).

SUMMARY:
The aim of this research is to evaluate thiol-disulfide balance in cervix cancer patients

DETAILED DESCRIPTION:
To date various oxidative stress parameters were studied in patients with cervix cancer, however dynamic thiol disulfide hemostasis has not been previously investigated.

The thiol-disulfide balance in the circulation will be measured by the automated system created by Erel & Neselioglu (1).

References

1- Erel O, Neselioglu S. A novel and automated assay for thiol/disulphide homeostasis. Clin Biochem 2014;47:326-32. doi:10.1016/j.clinbiochem.2014.09.026.

ELIGIBILITY:
Inclusion Criteria:

• Histopathologically confirmed diagnosis of cervix cancer

Exclusion Criteria:

* pulmonary disease
* pulmonary hypertension
* cardiac dysfunction
* renal dysfunction
* liver disease
* chronic ischemia
* systemic inflammation
* concomitant malignancy
* patients who use vitamin A,C or E (antioxidant vitamins)
* patients who use smoke
* patients who use drink alcohol
* patients who use addictive for any drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cervix cancer
Study Population: The preoperative diagnosis of cervix cancer was made histopathologically by cervical biopsy. An experienced pathologist performed pathological analysis according to the surgical staging scheme of the International Federation of Gynaecology and Obstetrics.
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
serum native thiol level | preoperative in the morning or preprandial for healthy volunteers
  serum native thiol level in μmol/L
serum disulphide level | preoperative in the morning or preprandial for healthy volunteers
  serum disulphide level in μmol/L
serum total thiol level | preoperative in the morning or preprandial for healthy volunteers
  serum total thiol level in μmol/L
the disulphide/native thiol ratio | preoperative in the morning or preprandial for healthy volunteers
  the disulphide/native thiol ratio X (100 )
disulphide/total thiol ratio | preoperative in the morning or preprandial for healthy volunteers
  disulphide/total thiol ratio X (100 )
native thiol/total thiol ratio | preoperative in the morning or preprandial for healthy volunteers
  native thiol/total thiol ratio X (100 )

SECONDARY OUTCOMES:
total oxidant capacity (TOC) | preoperative in the morning or preprandial for healthy volunteers
  TOC in mmol H2O2 equivalent/L
total antioxidant capacity (TAC) | preoperative in the morning or preprandial for healthy volunteers
  TAC in mmol trolox equivalent/L
Oxidative stress index (OSI) | preoperative in the morning or preprandial for healthy volunteers
  OSI in mmol trolox/L.
ischaemia-modified albumin | preoperative in the morning or preprandial for healthy volunteers
  ischaemia-modified albumin in IU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Burak Sezgin, MD, Principal Investigator — Mugla Sıtkı Kocman University Faculty of Medicine
Locations (1):
- Mugla Sıtkı Kocman University Faculty of Medicine, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided